CLINICAL TRIAL: NCT02232321
Title: Vascular Effects of Achieving Minimal Disease Activity in Psoriatic Arthritis - a 2 Year Prospective Cohort Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lai-Shan Tam, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PsA-MDA
Record Dates: First submitted 2014-09-02; First posted 2014-09-05 (Estimated); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Psoriatic Arthritis; Atherosclerosis; Arterial Stiffness
MeSH Terms: conditions — Arthritis, Psoriatic; Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PsA MDA (Other)
  Interventions: Other: PsA MDA

INTERVENTIONS:
Other: PsA MDA

SUMMARY:
Objectives To investigate the effect of achieving minimal disease activity (MDA) using a protocolized treatment strategy on the progression of subclinical atherosclerosis and arterial stiffness in psoriatic arthritis (PsA) patients.

Hypothesis Effective suppression of inflammation in patients who can achieve MDA will have less progression of subclinical atherosclerosis and arterial stiffness then patients who cannot achieve MDA by means of a standardized treatment algorithm aiming at MDA.

Design and subjects One hundred consecutive PsA patients will participate in this 2-year prospective, hospital-based, cohort study.

Interventions All participants will receive 2-year tight-control treatment. Treatment will be adjusted according to a standardized protocol based on the European League Against Rheumatism (EULAR) recommendation and the Hong Kong guideline on the use of biologics every 4-monthly aiming at MDA.

Study instruments Carotid intima-media thickness (IMT) will be measured using high-resolution ultrasound. Arterial stiffness is measured using pulse wave velocity (PWV) by a dedicated tonometry system and augmentation index (AIx) by the SphygmoCor device.

Main outcome measures and analysis The main outcome measure is the change in IMT over a period of 2 years comparing between patients who achieve MDA at 12 months (MDA group) to those who cannot achieve MDA (non-MDA group). Secondary outcomes include differences in the changes in AIx and PWV over 2 years between the 2 groups. Comparisons of the changes in IMT, AIx and PWV over 2 years between the MDA and non-MDA groups will be performed.

DETAILED DESCRIPTION:
Background:

Patients with psoriatic arthritis (PsA) experience substantial morbidity and unfavorable outcomes at referral centers. Although studies on all-cause mortality have yielded mixed results, increased cardiovascular (CV) mortality and morbidity in PsA have been consistently reported. Data from our group and others have shown that underlying these higher CV disease (CVD) rates is a greater burden of subclinical carotid atherosclerosis. Increased intima-media thickness (IMT) significantly correlates with traditional risk factors and disease-related parameters. An increased prevalence of arterial stiffness has also been demonstrated in patients with psoriasis and PsA compared with controls. In PsA, criteria for minimal disease activity (MDA) have been developed and validated. These criteria use 7 measurements including entheseal and skin assessments. Achieving MDA by these criteria results in less radiographic damage in the long term. The development of this instrument is a step toward 'treatment to target' in PsA. MDA is achieved in 48-60% of patients at ≥ 1 visit, and is sustained for ≥ 12 months (sustained MDA) in at least one third of PsA patients in a large observational cohort.

While achieving MDA may result in significant benefits in articular disease, little is known about its effect on extra-articular disease, including CVD risk. The use of surrogate end points instead of actual CV events may provide more evidence on whether PsA patients may benefit from potent anti-inflammatory treatment on the prevention of premature atherosclerosis. Data from our group and others linked the suppression of inflammation using anti-tumour necrosis factor (anti-TNF) with a favourable effect on CV surrogate makers, including carotid IMT and arterial stiffness. More recently, a tight-control treatment strategy aiming at remission was effective in improving arterial stiffness in our early rheumatoid arthritis (RA) cohort. There is an imperative need for interventional trials with CV end points to investigate whether achievement of MDA by a protocolized treatment strategy could reduce CVD risk in PsA. To fill in these gaps of knowledge, we propose a prospective cohort study to ascertain whether achieving MDA through a protocolized treatment strategy may prevent long term progression of IMT and arterial stiffness to a greater extent than those who cannot achieve MDA in patients with PsA.

Aim of the study:

Primary outcome:

1. Effect of achieving MDA (MDA group) at 12 months on the progression of subclinical atherosclerosis over a period of 24 months as evaluated by IMT compared to those who cannot achieve MDA (non-MDA group)

Secondary outcomes:

1. Changes in arterial stiffness over a period of 24 months as evaluated by pulse wave velocity (PWV) and augmentation Index (AIx) between the MDA group and non-MDA group.
2. The proportion of patients achieving sustained MDA (from 12 to 24 months)
3. Changes in IMT and arterial stiffness over a period of 24 months as evaluated by IMT, PWV and AIx between patients who can achieve sustained MDA and those who cannot achieve sustained MDA.
4. Correlations between the changes in IMT, PWV, and AIX and the changes in markers of disease activity

Hypothesis:

Effective suppression of inflammation in PsA patients who can achieve MDA will have less progression of subclinical atherosclerosis and arterial stiffness than patients who cannot achieve MDA by means of a protocolized treatment algorithm

ELIGIBILITY:
Inclusion Criteria:

* PsA attending the outpatient clinic of the Prince of Wales Hospital (PWH) who fulfilled the Classification of Psoriatic Arthritis criteria

Exclusion Criteria:

* 1) have a history of overt CVD (myocardial infarction, percutaneous transluminal coronary angioplasty, surgery for ischemic heart disease, stroke, transient ischemic attack, carotid endarterectomy, peripheral arterial reconstructive surgery, or limb amputation), or 2) are on aspirin, or HMG-CoA reductase inhibitors (statins) or angiotensin-converting-enzyme inhibitor (ACEI), or 3) have significant co-morbidities including severe renal impairment defined as a glomerular filtration rate of less than 30 mL/min/1.73m2, alanine aminotransferase (ALT) ≥2xULN, hemoglobin level <8.5gm/dl, white blood cell count <3.5x109/liter, platelet count<100x109/liter, or 4) female of childbearing potential who are unwilling to use adequate contraception, pregnant or breastfeeding women, or 5) they are on glucocorticoids at a dose >10mg/day (equivalent dose of prednisolone)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2014-03; Primary Completion 2017-10 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
PsA MDA and subclinical atherosclerosis | 30 months
  Effect of achieving MDA (MDA group) at 12 months on the progression of subclinical atherosclerosis over a period of 24 months as evaluated by IMT compared to those who cannot achieve MDA (non-MDA group).

SECONDARY OUTCOMES:
PsA MDA and arterial stiffness | 30 months
  Changes in arterial stiffness over a period of 24 months as evaluated by pulse wave velocity (PWV) and augmentation Index (AIx) between the MDA group and non-MDA group.
PsA MDA rate | 30 months
  The proportion of patients achieving sustained MDA (from 12 to 24 months)
PsA sustained MDA and atherosclerosis and arterial stiffness | 30 month
  Changes in IMT and arterial stiffness over a period of 24 months as evaluated by IMT, PWV and AIx between patients who can achieve sustained MDA and those who cannot achieve sustained MDA.
PsA atherosclerosis and arterial stiffness | 30 months
  Correlations between the changes in IMT, PWV, and AIX and the changes in markers of disease activity

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, China

REFERENCES:
- [Derived] Cheng IT, Shang Q, Li EK, Wong PC, Kun EW, Law MY, Yip RM, Yim IC, Lai BT, Ying SK, Kwok KY, Li M, Li TK, Zhu TY, Lee JJ, Chang MM, Szeto CC, Yan BP, Lee AP, Tam LS. Effect of Achieving Minimal Disease Activity on the Progression of Subclinical Atherosclerosis and Arterial Stiffness: A Prospective Cohort Study in Psoriatic Arthritis. Arthritis Rheumatol. 2019 Feb;71(2):271-280. doi: 10.1002/art.40695. Epub 2019 Jan 5. PMID 30144299
- [Derived] Shen J, Wong KT, Cheng IT, Shang Q, Li EK, Wong P, Kun EW, Law MY, Yip R, Yim I, Ying S, Li M, Li TK, Wong CK, Zhu TY, Lee JJ, Chang M, Lee AP, Tam LS. Increased prevalence of coronary plaque in patients with psoriatic arthritis without prior diagnosis of coronary artery disease. Ann Rheum Dis. 2017 Jul;76(7):1237-1244. doi: 10.1136/annrheumdis-2016-210390. Epub 2017 Jan 4. PMID 28052860